CLINICAL TRIAL: NCT07097636
Title: Effect of Video Education on Anxiety and Satisfaction Levels of Parents of Children Undergoing Urodynamic Studies
Acronym: Video Educatio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Rüya Naz, Principal Investigator, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2011-KAEK-25 2023/07-09
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Satisfaction
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention (Experimental): Video education
  Interventions: Other: Video education
- No intervention (Other): Control group
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Video education — A video demonstrating the steps of the urodynamic procedure was shown, and afterward, participants' questions were answered by an experienced nurse who performed the procedure.
  Other Names: İntervention group
  Arms: İntervention
Other: No intervention — Children scheduled to undergo urodynamic testing for any reason received the procedure without any prior video-based education being provided to their parents
  Other Names: Control group
  Arms: No intervention

SUMMARY:
The aim of this study was to evaluate the effects of video-based education provided to parents of children undergoing urodynamic testing on their State-Trait Anxiety Inventory and satisfaction levels. While some of the parents of children scheduled for urodynamic testing were shown a video, others were not. Anxiety and satisfaction levels were assessed in both groups before and after the procedure.

DETAILED DESCRIPTION:
This study was conducted at Bursa Yuksek Ihtisas Training and Research Hospital between July 2023 and January 2024 to evaluate the effect of video-based education provided to parents of children undergoing urodynamic testing on their anxiety and satisfaction levels. Participants were randomly assigned to two groups. In the control group, parents received information about the urodynamic procedure from the nurses performing the test. In the intervention group, in addition to receiving information, the parents were shown a video explaining the urodynamic procedure. All questions from the participants were answered by the nurse conducting the urodynamic procedure. A total of 140 patients were planned to be included in the study, with 70 in each group. The State-Trait Anxiety Inventory (STAI) was used to assess anxiety levels, and a verbal descriptive scale was used to evaluate satisfaction with the procedure.

ELIGIBILITY:
Inclusion Criteria:Parents must be at least 18 years old,

* Parents must be at least 18 years old
* have no intellectual disabilities or perception problems
* have no communication difficulties.

Exclusion Criteria

* Insufficient proficiency in Turkish and unwillingness to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Parents' anxiety levels before the education | Immediately before procedurel]
  Anxiety levels before the procedure will be assessed using the State-Trait Anxiety Inventory, which consists of 20 questions. Each question is scored from 1 to 4. A total score below 30 indicates low anxiety, a score between 31 and 45 indicates moderate anxiety, and a score of 46 or above indicates high anxiety. The urodynamic procedure will be performed according to routine clinical practice. High scores indicate high anxiety, while low scores indicate low anxiety.
Parents' anxiety levels after the education | Immediately after education
  Parents in the control group will receive only verbal information, while parents in the study group will be given verbal education as well as shown a video. After the education, the anxiety levels of the parents will be assessed using the State-Trait Anxiety Inventory - State (STAI-S).

SECONDARY OUTCOMES:
Parental satisfaction levels regarding the video training | Immediately after the education
  The satisfaction levels of parents in the intervention group after the video training were evaluated using a verbal descriptive scale. This scale is rated as follows:
  I) Not satisfied at all II) Not satisfied III) Neither satisfied nor dissatisfied IV) Satisfied V) Very satisfied High scores indicate high satisfaction, while low scores indicate low satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yüksek İhtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 6 month